CLINICAL TRIAL: NCT03061370
Title: An Investigation of the Prevalence and Clinical Impact of Sarcopenia and Visceral Obesity Among Patients With Upper Gastrointestinal Malignancies
Brief Title: Sarcopenia and Visceral Obesity in Esophageal and Gastric Cancer
Status: Completed | Type: Observational
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Clinical Research Fellow, St. James's Hospital, Ireland
Other Study IDs: SJHDOS2016-01
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Cancer; Gastric Cancer; Sarcopenia; Sarcopenic Obesity; Obesity; Visceral Obesity; Quality of Life; Surgery; Complication of Treatment; Chemotherapeutic Toxicity; Physical Activity; Oncology
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Sarcopenia; Obesity; Obesity, Abdominal; Motor Activity; Neoplasms | interventions — Esophagectomy; Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Esophagectomy or Gastrectomy — Surgical resection

SUMMARY:
In line with improvements in oncologic outcome for patients with esophageal cancer, the attritional impact of curative treatment with respect to functional status and health-related quality of life (HR-QL) in survivorship is increasingly an important focus. Functional recovery after surgery for esophageal cancer is commonly confounded by anorexia and early satiety, which may reduce oral nutrient intake with consequent malnutrition and weight loss. One in three disease-free patients has more than fifteen percent body weight loss at three years after esophagectomy.

The ESPEN Special Interest Group on cachexia-anorexia in chronic wasting diseases has defined sarcopenia as skeletal muscle index (SMI) of ≤39 cm2/m2 for women and ≤55cm2/m2 for men, while similar cut-off points have been validated in upper gastrointestinal and respiratory malignancies (less than 38.5 cm2/m2 for women and 52.4 cm2/m2 for men). The European Working Group on Sarcopenia in Older People (EWGSOP) additionally recommends that assessment should also include determination of muscle function, for example gait speed or grip strength, where possible.

The presence of sarcopenia is associated with increase treatment-associated morbidity, impaired HR-QL, reduced physical and role functioning, and increased pain scores in older adults. In addition, a previous longitudinal study demonstrated that the decline in HR-QL over a six year period in older adults was accelerated in the presence of sarcopenia. As such, sarcopenia may represent a modifiable barrier to recovery and subsequent retention of HR-QL and functional status, and may reinforce a persistent illness identity, among patients following potentially curative treatment for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Initial staging computed tomography (CT) scan capturing the level of the L3 conducted at our Centre and available for review

Exclusion Criteria:

* Patients who had a history of previous gastrointestinal resection, other active malignancy, eating disorder, inflammatory bowel disease or other significant illness that might alter body composition were excluded from analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal or gastric cancer between 2010 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Neoadjuvant therapy toxicity | 6 months
Postoperative morbidity | 6 months
Oncologic outcome | 6 months
Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John V Reynolds, MCh FRCS, Principal Investigator — Department of Surgery, St. James's Hospital, Dublin
Locations (2):
- Ireland (2):
  - Department of Surgery, St. James's Hospital, Dublin
  - Wellcome Trust-Health Research Board Clinical Research Facility, St. James's Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prado CM, Lieffers JR, McCargar LJ, Reiman T, Sawyer MB, Martin L, Baracos VE. Prevalence and clinical implications of sarcopenic obesity in patients with solid tumours of the respiratory and gastrointestinal tracts: a population-based study. Lancet Oncol. 2008 Jul;9(7):629-35. doi: 10.1016/S1470-2045(08)70153-0. Epub 2008 Jun 6. PMID 18539529
- [Background] Doyle SL, Bennett AM, Donohoe CL, Mongan AM, Howard JM, Lithander FE, Pidgeon GP, Reynolds JV, Lysaght J. Establishing computed tomography-defined visceral fat area thresholds for use in obesity-related cancer research. Nutr Res. 2013 Mar;33(3):171-9. doi: 10.1016/j.nutres.2012.12.007. Epub 2013 Jan 30. PMID 23507222
- [Result] Elliott JA, Doyle SL, Murphy CF, King S, Guinan EM, Beddy P, Ravi N, Reynolds JV. Sarcopenia: Prevalence, and Impact on Operative and Oncologic Outcomes in the Multimodal Management of Locally Advanced Esophageal Cancer. Ann Surg. 2017 Nov;266(5):822-830. doi: 10.1097/SLA.0000000000002398. PMID 28796017